CLINICAL TRIAL: NCT03479164
Title: Development of Ultra-Low Dose CT Based Screening for Aortic Aneurysms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1510M79442
Record Dates: First submitted 2018-03-07; First posted 2018-03-27 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Aortic Aneurysm, Thoracic; Aortic Aneurysm, Abdominal
MeSH Terms: conditions — Aortic Aneurysm, Thoracic; Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultra Low-Dose CT (Experimental): One non-contrast gated aortic (NCGA) computer tomography scan, a low radiation, non-contrast, low cost CT based study
  Interventions: Other: Ultra Low-Dose CT

INTERVENTIONS:
Other: Ultra Low-Dose CT — Ultra Low-Dose CT

SUMMARY:
The primary objective of this research project is development and validation of a new, non-contrast gated aortic (NCGA) computer tomography scan algorithm for screening of aortic aneurysm in the chest and abdomen in at risk patients. This study would initially be performed in patients with a known aneurysm and done in addition to their indicated surveillance CT scan.

DETAILED DESCRIPTION:
Study Design: Patients who agree to enroll in the study will get the NCGA study as well as a routine non-contrast computed tomography of chest/abdomen/pelvis within one year following recruitment at the patient's convenience. No follow-up will be required, but any clinically relevant findings on the testing will be communicated to the PCP through EPIC in-basket. Urgent findings, as determined by the primary investigator, will also result in a direct communication with the PCP. It is expected that any such findings will also be seen on the standard and clinically indicated CT which they are also undergoing, and so "new or unique" findings on the study NCGA test are not expected to occur. The final study visit will be the day of participation.

Study Design: Patients who agree to enroll in the study will get the NCGA study as well as a routine non-contrast computed tomography of chest/abdomen/pelvis within one year following recruitment at the patient's convenience. No follow-up will be required, but any clinically relevant findings on the testing will be communicated to the PCP through EPIC in-basket. Urgent findings, as determined by the primary investigator, will also result in a direct communication with the PCP. It is expected that any such findings will also be seen on the standard and clinically indicated CT which they are also undergoing, and so "new or unique" findings on the study NCGA test are not expected to occur. The final study visit will be the day of participation.

Study Procedures: One visit to complete one (1) non-contrast (no "dye"/contrast material will be injected) computed tomography (CT) scan of the chest, abdomen and pelvis. This visit will occur within one year following recruitment, scheduled at the patient's convenience. This one visit represents the totality of study participation for each participant.

Study Duration: For each individual, participation is only over one day - the day of the patient's non-contrast CT scan. No early termination visits or unscheduled visits apply.

The anticipated duration to complete enrollment of all participants is 1 year. Following completion of the study, the study team is planning for an interim period of 6 months for discussion and planning for future projects.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who carry the diagnosis of thoracic aortic aneurysm, aortic dissection, or abdominal aortic aneurysm and require CT imaging to evaluate the pathology

Exclusion Criteria:

* Current pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-03-30 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Effectiveness of Ultra Low-Dose CT | Day of Scan
  To assess the sensitivity of NCGA for aortic aneurysm in the thoracic or abdominal aorta

SECONDARY OUTCOMES:
Radiation Exposure of Ultra Low-Dose CT | Day of Scan
  To assess the relative radiation exposure of NCGA to the patient in comparison to a standard CT

OTHER OUTCOMES:
Assess Findings of Ultra Low-Dose CT | Day of Scan
  To assess the success of limiting extraneous findings of the test.
Optimize Automation of Ultra Low-Dose CT | Day of Scan
  To optimize automation of the test.

CONTACTS AND LOCATIONS:
Overall Officials: Rumi Faizer, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota - Twin Cities, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No